CLINICAL TRIAL: NCT04670874
Title: Assessment of Quality of Life in Cutaneous Lymphoma Patients Using the Skindex29
Brief Title: Quality of Life in Cutaneous Lymphoma Patients Using the Skindex29
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22364; NCI-2020-11058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22364 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (quality of life questionnaire): Patients complete quality of life questionnaires over 10-20 minutes about symptoms, emotions, and functioning related to diagnosis of cutaneous lymphoma.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete quality of life questionnaire
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete quality of life questionnaire

SUMMARY:
This study assesses the quality of life in patients with cutaneous lymphoma diagnosis as it relates to their personal, clinical, and therapeutic information using the Skindex29 questionnaire and also assesses patients' understanding of their diagnosis and need for resources related to their care. Cutaneous lymphomas are a rare type of blood cancers (non-Hodgkin lymphoma) that present in the skin. The information gained from this study, may help researchers improve quality of life in cutaneous lymphoma patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively assess quality of life (QoL) in adult patients with cutaneous lymphoma (CL) via use of a validated questionnaire (Skindex-29) and identify the psychosocial needs of our patient population.

II. To prospectively evaluate the burden of pruritus in patients with CL via use of 10-point pruritus scale and compare to QoL.

III. To evaluate QoL for any correlation with demographic and clinical information, specifically, age, gender, race/ethnicity, type of CL, stage of mycosis fungoides (MF)/Sezary syndrome (SS), treatment regimen, and social work involvement.

IV. To track changes in QoL and burden of pruritus as they relate to therapeutic strategies used to manage disease, including social work involvement.

V. To prospectively assess patients' knowledge and understanding of their cancer diagnosis, prognosis, and overall survival; and to track changes in their knowledge and understanding, and assess for any correlation to QoL.

VI. To prospectively evaluate our patients' need for resources, and our ability to meet those needs; and to assess for any correlation to demographic or clinical category, or QoL.

OUTLINE:

Patients complete quality of life questionnaires over 10-20 minutes about symptoms, emotions, and functioning related to diagnosis of cutaneous lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the research study
* Presumed or confirmed diagnosis of CL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with presumed or confirmed diagnosis of CL who present to the Multidisciplinary CL Clinic at City of Hope
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2034-01-24 (Estimated); Study Completion 2034-01-24 (Estimated)

PRIMARY OUTCOMES:
Skindex-29 domain (symptom, function, and emotion) scores | At completion of questionnaire
  Skindex-29 domain (symptom, function, and emotion) scores will be summarized by diagnosis group, demographics, disease characteristics, treatment/intervention, and disease response/clinical outcome. Cross-sectional and longitudinal summary of the data will be performed. Descriptive statistics for continuous data (mean, standard deviation, median, range, etc.) will be used to summarize quality of life. Descriptive and summary statistics or continuous and categorical data (counts and percentages) will be used to summarize continuous or categorical demographics or other patient/disease characteristics respectively. Graphical representation of the data will be used when helpful. Descriptive statistics for categorical data will be used to assess patients' understanding of their cancer diagnosis and need for resources based on the survey.
Burden of pruritus | At completion of questionnaire
  Burden of pruritus as measured by pruritus scale will be summarized by diagnosis group, demographics, disease characteristics, treatment/intervention, and disease response/clinical outcome. Cross-sectional and longitudinal summary of the data will be performed. Descriptive statistics for continuous data (mean, standard deviation, median, range, etc.) will be used to summarize pruritus score. Descriptive and summary statistics or continuous and categorical data (counts and percentages) will be used to summarize continuous or categorical demographics or other patient/disease characteristics respectively. Graphical representation of the data will be used when helpful. Descriptive statistics for categorical data will be used to assess patients' understanding of their cancer diagnosis and need for resources based on the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Querfeld, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States